CLINICAL TRIAL: NCT01990781
Title: Combined Effect of Intravenous Lidocaine and Dexamethasone on Postoperative Sore Throat, Cough and Hoarseness. A Randomized Controlled Trial
Brief Title: Effect of Intravenous Lidocaine and Dexamethasone Combination on Postoperative Sore Throat, Cough and Hoarseness.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Asish Subedi, Associate Professor, Department of Anesthesiology, BPKIHS, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 387/070/071
Record Dates: First submitted 2013-11-02; First posted 2013-11-21 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Postoperative Sore Throat, Cough, Hoarseness
Keywords: Lidocaine, Dexamethasone, Postoperative sore throat
MeSH Terms: conditions — Cough; Hoarseness | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group LD: Lidocaine and Dexamethasone (Experimental): lidocaine 1.5 mg/kg and dexamethasone (dexona) 8 mg iv prior to induction of anesthesia
  Interventions: Drug: LD: Lidocaine and dexamethasone
- Group L: Lidocaine (Active Comparator): Group L: lidocaine 1.5 mg/kg iv prior to induction of anesthesia
  Interventions: Drug: L:Lidocaine
- D: Dexamethasone (Active Comparator): Dexamethasone 8 mg iv prior to induction of anesthesia
  Interventions: Drug: D: Dexamethasone
- N: normal saline (Placebo Comparator): N: normal saline (placebo): 2 ml
  Interventions: Drug: N: Normal saline (placebo)

INTERVENTIONS:
Drug: LD: Lidocaine and dexamethasone — LD: intravenous lidocaine 1.5 mg/kg and dexamethasone 8 mg before induction of anesthesia
  Other Names: Xylocard, dexona
  Arms: Group LD: Lidocaine and Dexamethasone
Drug: L:Lidocaine — Intravenous lidocaine 1.5 mg/kg before induction of anesthesia
  Other Names: Xylocard
  Arms: Group L: Lidocaine
Drug: D: Dexamethasone — D:intravenous dexamethasone 8 mg before induction of anesthesia
  Other Names: Dexona
  Arms: D: Dexamethasone
Drug: N: Normal saline (placebo) — Normal saline: 2ml
  Arms: N: normal saline

SUMMARY:
Post operative sore throat (POST) following tracheal intubation is a common problem causing dissatisfaction and discomfort to the patients. Prophylactic use of both lidocaine and dexamethasone has been used independently for this purpose. However, there is no study assessing the synergistic analgesic effects of lidocaine and dexamethasone for POST. The purpose of this study is to compare the effect of lidocaine, dexamethasone and lidocaine dexamethasone combination on the incidence and severity of POST.

DETAILED DESCRIPTION:
Sore throat and hoarseness following tracheal intubation are common postoperative problems causing dissatisfaction and discomfort to the patients. Their incidence varies from 30%-70%.

Both non pharmacological and pharmacological measures have been tried to minimize the incidence and severity of POST with variable success rate. Prophylactic use lidocaine and steroids have been used independently for this purpose. Dexamethasone as an adjuvant to lidocaine has shown to improve the quality of analgesia. However, there is no study assessing the combine effects of lidocaine and dexamethasone for POST.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologist(ASA) physical status 1 & 2 requiring general anesthesia with endotracheal intubation.
* Duration of surgery more than 90 min

Exclusion Criteria:

* Those with preexisting hoarseness or sorethroat
* Smoker
* Vocal performer by occupation
* Recent or recurrent respiratory tract infection
* Risk factors for postoperative aspiration
* Obesity
* Pregnancy
* Receiving analgesics, corticosteroids and calcium channel blockers
* Contraindication to corticosteroid medications
* Anticipated difficult intubation
* Mallampati grade > 2
* Difficult mask ventilation requiring oral or nasal airway
* Cormack and Lehman grade III and IV on laryngoscopy
* More than one intubation attempt
* Those requiring orogastric or nasogastric tubes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative sore throat at rest and on swallowing. | From 1 to 24 hr following surgery
  Incidence of postoperative sore throat. Assessment of severity of postoperative sorethroat using scoring system, 0-No sore throat at any time since the operation,1- Minimal sore throat,2- Moderate sore throat,3- Severe sore throat

SECONDARY OUTCOMES:
-Assessment of post operative cough. Assessment of post operative cough using scoring system,0- No cough,1- Minimal cough,2- Moderate cough,3- Severe cough. | From 1 to 24 hr following surgery
  -Assessment of postoperative hoarseness. Assessment of postoperative hoarseness using scoring system,0- No evidence of hoarseness at any time since the operation,1-No evidence of hoarseness at the time of interview,2-Hoarseness at the time of interview noted by patient only, 3- Hoarseness that is easily noted at the time of interview

CONTACTS AND LOCATIONS:
Overall Officials: Asish Subedi, MD, Principal Investigator — BPKIHS
Locations (1):
- BP Koirala Institute of Health Sciences (BPKIHS), Dharān, Koshi, Nepal

REFERENCES:
- [Derived] Subedi A, Tripathi M, Pokharel K, Khatiwada S. Effect of Intravenous Lidocaine, Dexamethasone, and Their Combination on Postoperative Sore Throat: A Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):220-225. doi: 10.1213/ANE.0000000000003842. PMID 30320641